CLINICAL TRIAL: NCT05288075
Title: Pharmacokinetic Formulation Feasibility Study to Compare Relative Bioavailability of 3 Indacaterol/Glycopyrronium Easyhaler Test Products and Reference Product Ultibro Breezhaler
Brief Title: Study to Compare Relative Bioavailability of 3 Indacaterol/Glycopyrronium Test Products and Reference Product
Acronym: FORELLI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3131002
Record Dates: First submitted 2022-02-07; First posted 2022-03-18 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — indacaterol; Glycopyrrolate; Charcoal; Hardness

STUDY DESIGN:
Masking Description: Bioanalytical laboratory will be blinded with regard to the sequence of the product administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Indacaterol/glycopyrronium Easyhaler® 85/43 µg/dose, inhalation powder, product variant A (Experimental): Each subject will receive a single dose of 2 inhaled doses from Indacaterol/glycopyrronium Easyhaler product variant A in one of the four periods (cross-over) with concomitant charcoal administration (Carbomix granules). The total dose is 170 µg of indacaterol and 86 µg glycopyrronium (delivered doses).
  Interventions: Drug: Indacaterol/glycopyrronium
- Indacaterol/glycopyrronium Easyhaler® 85/43 µg/dose, inhalation powder, product variant B (Experimental): Each subject will receive a single dose of 2 inhaled doses from Indacaterol/glycopyrronium Easyhaler product variant B in one of the four periods (cross-over) with concomitant charcoal administration (Carbomix granules). The total dose is 170 µg of indacaterol and 86 µg glycopyrronium (delivered doses).
  Interventions: Drug: Indacaterol/glycopyrronium
- Indacaterol/glycopyrronium Easyhaler® 85/43 µg/dose, inhalation powder, product variant C (Experimental): Each subject will receive a single dose of 2 inhaled doses from Indacaterol/glycopyrronium Easyhaler product variant C in one of the four periods (cross-over) with concomitant charcoal administration (Carbomix granules). The total dose is 170 µg of indacaterol and 86 µg glycopyrronium (delivered doses).
  Interventions: Drug: Indacaterol/glycopyrronium
- Ultibro® Breezhaler® 85/43 µg inhalation powder, hard capsule (Active Comparator): Each subject will receive 2 capsules of Ultibro® Breezhaler® (=Indacaterol/glycopyrronium) as a single dose in one of the four periods (cross-over) with concomitant charcoal administration (Carbomix granules). The total dose is 170 µg of indacaterol and 86 µg glycopyrronium (delivered doses).
  Interventions: Drug: Indacaterol/glycopyrronium

INTERVENTIONS:
Drug: Indacaterol/glycopyrronium — In each period, subjects receive single dose of indacaterol/glycopyrronium consisting of 2 inhaled doses via Easyhaler or 2 capsules inhaled via Ultibro Breezhaler.
  In addition to study treatments, activated charcoal will be administered on each study period before and after study drug administration.
  Other Names: Indacaterol/glycopyrronium Easyhaler® 85/43 µg/dose, inhalation powder, product variant A with charcoal; Indacaterol/glycopyrronium Easyhaler® 85/43 µg/dose, inhalation powder, product variant B with charcoal; Indacaterol/glycopyrronium Easyhaler® 85/43 µg/dose, inhalation powder, product variant C with charcoal; Ultibro® Breezhaler® 85/43 µg inhalation powder, hard capsule with charcoal

SUMMARY:
This is a formulation feasibility study to to compare relative bioavailability of indacaterol and glycopyrronium after administration of single doses of 3 Easyhaler test products and Ultibro Breezhaler. The study treatments will be administered with concomitant oral charcoal to block absorption via gastrointestinal tract and to assess pulmonary absorption only.

ELIGIBILITY:
Main Inclusion Criteria:

1. Healthy males and females
2. 18-60 years of age
3. Body mass index 19-30 kg/m2
4. Weight at least 50 kg
5. Written informed consent obtained

Main Exclusion Criteria:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, GI, pulmonary, metabolic, endocrine, neurological or psychiatric disease
2. Any condition requiring regular concomitant treatment
3. Any clinically significant abnormal laboratory value, vital sign or physical finding that in the opinion of the investigator could interfere with the interpretation of study results or cause a health risk for the subject
4. Known hypersensitivity to indacaterol or glycopyrronium
5. Pregnant or lactating females and females of childbearing potential not using contraception of acceptable effectiveness
6. Blood donation or loss of significant amount of blood within 90 days prior to the first study treatment administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Peak indacaterol and glycopyrronium concentration in plasma (Cmax) | between 0-72 hours after dosing
  Pharmacokinetic parameters of indacaterol and glycopyrronium
Area under the concentration-time curve from time zero to 72 hours (AUC72) | between 0-72 hours after dosing
  Pharmacokinetic parameters of indacaterol and glycopyrronium

SECONDARY OUTCOMES:
Time to reach peak indacaterol and glycopyrronium concentration in plasma (tmax) | between 0-72 hours after dosing
  Pharmacokinetic parameters of indacaterol and glycopyrronium
Area under the concentration-time curve from time zero to 30 minutes (AUC30) | between 0-30 minutes after dosing
  Pharmacokinetic parameters of indacaterol and glycopyrronium

OTHER OUTCOMES:
Adverse events | Up to 11 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Orion Corporation Clinical Study Director, Study Director — Orion Corporation, Orion Pharma; Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- CRST Helsinki Oy, Helsinki, Finland